CLINICAL TRIAL: NCT01578356
Title: Oncological and Functional Outcomes After Radical Prostatectomy for Prostate Cancer: Comparing Open With Robot-assisted Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/122
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Radical Retropubic prostatectomy (RRP): Men who underwent open radical prostatectomy in the past at our centre.
- Robot-assisted laparoscopic prostatectomy (RALP): Men who undergo robot-assisted laparoscopic prostatectomy at our centre.

SUMMARY:
For primary surgical treatment of prostate cancer the investigators compare the classic open surgery (radical retropubic prostatectomy, RRP) versus robot-assisted laparoscopic surgery (RALP). Oncological results are obtained at standard follow-up consultations through Prostate-Specific Antigen (PSA) measurement to detect biochemical recurrence. Functional results (continence, potency, quality of life) are obtained through standardised questionnaires. Currently the investigators perform all of their prostatectomies in a robot-assisted manner. For results of the open surgery the investigators send questionnaires to patients who had the operation in the past.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer
* radical retropubic prostatectomy or
* robot-assisted laparoscopic surgery

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who were surgically treated or who are being surgically treated for prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2011-10-31 (Actual); Study Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
Biochemical recurrence at follow-up. | 3 months after prostatectomy
  PSA measurement in the serum should not be > or = 0,20 ng/ml.
Biochemical recurrence at follow-up | 6 months after prostatectomy
  PSA measurement in the serum should not be > or = 0,20 ng/ml.
Biochemical recurrence at follow-up. | 9 months after prostatectomy
  PSA measurement in the serum should not be > or = 0,20 ng/ml.
Biochemical recurrence at follow-up. | 1 year after prostatectomy
  PSA measurement in the serum should not be > or = 0,20 ng/ml.
Biochemical recurrence at follow-up. | 6-monthly follow up between 1 and 5 years after prostatectomy.
  PSA measurement in the serum should not be > or = 0,20 ng/ml.

SECONDARY OUTCOMES:
Functional assessment concerning continence. | after 1, 3, 12 and 24 months
  Patients need to fill out questionnaires (EORTC QLQ-C30, QLQ-PR25, ICIQ mLUTS and UI SF and IIEF). The patients in the radical retropubic prostatectomy group only fill out the questionnaires once.
Functional assessment concerning potency. | after 1, 3, 12 and 24 months
  Patients need to fill out questionnaires (EORTC QLQ-C30, QLQ-PR25, ICIQ mLUTS and UI SF and IIEF). The patients in the radical retropubic prostatectomy group only fill out the questionnaires once.
Functional assessment concerning quality of life. | after 1, 3, 12 and 24 months
  Patients need to fill out questionnaires (EORTC QLQ-C30, QLQ-PR25, ICIQ mLUTS and UI SF and IIEF). The patients in the radical retropubic prostatectomy group only fill out the questionnaires once.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be